CLINICAL TRIAL: NCT03765060
Title: Clinical Trial on the Efficacy and Security of the Small Stitch Technique Versus the Large Stitch Closure Laparotomy Technique in Emergency Surgery
Brief Title: The Efficacy and Security of the Small Stitch Technique in Emergency Surgery
Acronym: STCU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SL-Stitch
Record Dates: First submitted 2018-08-08; First posted 2018-12-05 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Abdominal Wall Defect; Abdominal Wall Hernia; Eventration; Evisceration; Operation Wound
MeSH Terms: conditions — Hernia, Abdominal; Gastroschisis | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Stitch (Experimental): Patients requiring an urgent emergency laparotomy. The Small Stitch closure technique will be perform using a Monomax® 2/0 HR26 (Half-circle Round body):
  * It will be use a very long-term monofilament absorbable synthetic suture of Poly-4-hydroxybutyrate (Monomax) 2/0 with HR 26 needle (Half-circle Round body).
  * In the technique should be given at least 2 points for each wound cm, with a distance to the alba line of 0'5cm and 0'5 cm of separation between stitches. The closure starts from both ends, ending in the middle of the laparotomy with an overlap of at least 2 cm. The ratio between the length of the suture and the length of the wound should be at least 4:1.
  Interventions: Procedure: Monomax® 2/0 HR26
- Large Stitch (Active Comparator): The intervention will be the classic large Stitch closure technique using a Monomax® 1 HR48 (Half-circle Round body).
  * It will be use a very long-term monofilament absorbable synthetic suture of Poly-4-hydroxybutyrate (Monomax) 1 with HR 48 needle (Half-circle Round body).
  * In the technique should be given 1 point for each wound cm, with a distance to the alba line of 1 cm and 1 cm of separation between stitches. The closure starts from both ends, ending in the middle of the laparotomy with an overlap of at least 2 cm. The ratio between the length of the suture and the length of the wound should be at least 4:1.
  Interventions: Procedure: Monomax® 1 HR48

INTERVENTIONS:
Procedure: Monomax® 2/0 HR26 — It will be use a very long-term monofilament absorbable synthetic suture of Poly-4-hydroxybutyrate (Monomax) 2/0 with HR 26 needle.
  In the technique should be given at least 2 points for each wound cm, with a distance to the alba line of 0'5cm and 0'5 cm of separation between stitches. The closure starts from both ends, ending in the middle of the laparotomy with an overlap of at least 2 cm. The ratio between the length of the suture and the length of the wound should be at least 4:1.
  Other Names: Suture
  Arms: Small Stitch
Procedure: Monomax® 1 HR48 — It will be use a very long-term monofilament absorbable synthetic suture of Poly-4-hydroxybutyrate (Monomax) 1 with HR 48 needle.
  In the technique should be given 1 point for each wound cm, with a distance to the alba line of 1 cm and 1 cm of separation between stitches. The closure starts from both ends, ending in the middle of the laparotomy with an overlap of at least 2 cm. The ratio between the length of the suture and the length of the wound should be at least 4:1.
  Other Names: Suture
  Arms: Large Stitch

SUMMARY:
This study evaluates the abdominal closure technique in emergency surgery. Half of participants will be perform the classic Large Stitch technique, while the other half will undergo the Small Stitch technique.

DETAILED DESCRIPTION:
The closure of laparotomy is one of the most important challenges facing the surgeon.

The classic technique of wall closure is the Large Stitch technique that uses monofilament double-strand sutures with a SL/WL (Suture Lengh/Wound Lengh) 4:1 ratio, with a distance to the alba line and between each stitch of 1 cm.

Nowadays, the Small Stitch technique is accepted as the technique of choice for closure of laparotomies in programmed surgery. It is based on a very long-term monofilament absorbable synthetic suture of Poly-4-hydroxybutyrate (Monomax) 2/0 with HR (Half-circle Round body) 26 needle. Stitches should be given with a distance to the alba line of 0'5cm and 0'5 cm of separation between stitches.

There are very few studies about the role of Small Stitch technique in the field of Emergency Surgery where the increased morbidity of the patient and the higher rate of surgical wound infection can play a fundamental role, and could be improved with the use of new abdominal wall closure techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age and who provide informed consent to participate in the study.
2. Patients requiring an urgent midline laparotomy with a minimum size of 8 cm.

Exclusion Criteria:

1. Prior midline laparotomy.
2. Patients with BMI> 45 kg / m2
3. Patients with ASA (American Society of Anesthesiologists)> IV.
4. Patient with an advanced terminal illness with an expectation of life <1 year.
5. Patients with abdominal aortic aneurysm.
6. Patients with coagulopathy: patient previously diagnosed with von Willebrand disease, hemophilia or Immune thrombocytopenic purpura.
7. Immunosuppressed patient: HIV patients in the AIDS phase, chronic corticosteroid or immunosuppressive treatment.
8. Patients with collagen pathology: patient previously diagnosed with Marfan syndrome, Ehlers-Danlos syndrome, homocystinuria and scleroderma.
9. Chemotherapeutic treatment 2 weeks before surgery.
10. Radiotherapy treatment 6 weeks before surgery.
11. Diffuse peritonitis with hemodynamic instability, defined by non-response to fluids prior to surgery or during the surgical process.
12. Pregnant or potentially fertile women, breastfeeding, or intention to become pregnant, or those who do not wish to use effective contraception (hormonal contraceptives (implantation, patches, oral), and double barrier methods (any double combination of: IUD (intrauterine device), male or female prophylactics with spermicidal gel, diaphragm, contraceptive sponge, cervical cap).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the small stitch technique defined by eventration rate | 1 year
  To determine the efficacy of the "Small stitch" technique versus the "Large Stitch" technique in the closure of midline laparotomy with respect to the production of eventration in patients undergoing urgent abdominal surgery.

SECONDARY OUTCOMES:
Efficacy of the small stitch technique defined by local complications rate | 1 year
  To determine whether the closure of midline laparotomy with the "Small Stitch" technique in patients undergoing urgent abdominal surgery reduces the local complications of the surgical wound defined by hematoma, seroma or wound infection.
Efficacy of the small stitch technique defined by evisceration rate | 1 year
  To determine if the closure of the midline laparotomy with the "Small Stitch" technique in patients undergoing urgent abdominal surgery reduces the rate of evisceration.
Efficacy of the small stitch technique defined by improvement of quality of life | 1 year
  To determine if the closure of a midline laparotomy with the "Small Stitch" technique in patients undergoing urgent abdominal surgery improves the quality of life.
Security of the small stitch technique | 1 year
  To determine the safety of the Small Stitch technique versus the "Large Stitch" technique in the closure of the midline laparotomy with respect to the incidence of adverse events and serious adverse events, the incidence of side effects related to the treatment and the incidence and the reasons for premature withdrawal of premature patient from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tamayo López María Jesús, PhD, Principal Investigator — Hospital Universitario Virgen del Rocio; Padillo Ruiz Francisco Javier, PhD, Study Director — Hospital Universitario Virgen del Rocio
Locations (1):
- Hospital Universitario Virgen Del Rocio, Seville, Spain

REFERENCES:
- [Background] Israelsson LA, Millbourn D. Closing midline abdominal incisions. Langenbecks Arch Surg. 2012 Dec;397(8):1201-7. doi: 10.1007/s00423-012-1019-4. Epub 2012 Nov 11. PMID 23143146
- [Background] Millbourn D, Cengiz Y, Israelsson LA. Risk factors for wound complications in midline abdominal incisions related to the size of stitches. Hernia. 2011 Jun;15(3):261-6. doi: 10.1007/s10029-010-0775-8. Epub 2011 Jan 30. PMID 21279664
- [Background] Millbourn D, Wimo A, Israelsson LA. Cost analysis of the use of small stitches when closing midline abdominal incisions. Hernia. 2014;18(6):775-80. doi: 10.1007/s10029-013-1135-2. Epub 2013 Jul 10. PMID 23839330
- [Background] O'Dwyer PJ, Courtney CA. Factors involved in abdominal wall closure and subsequent incisional hernia. Surgeon. 2003 Feb;1(1):17-22. doi: 10.1016/s1479-666x(03)80004-5. PMID 15568420
- [Background] Israelsson LA, Jonsson T. Suture length to wound length ratio and healing of midline laparotomy incisions. Br J Surg. 1993 Oct;80(10):1284-6. doi: 10.1002/bjs.1800801020. PMID 8242299